CLINICAL TRIAL: NCT05709067
Title: Probiotics Effect on Mental Wellness
Acronym: Moa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fonterra Research Centre (Industry)
Collaborators: Sun Genomics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Moa
Record Dates: First submitted 2022-12-19; First posted 2023-02-01 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Mental Health Wellness
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Arm (Experimental)
  Interventions: Dietary Supplement: Probiotic
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — 6 Billion CFU per day
  Arms: Probiotic Arm
Dietary Supplement: Placebo — 0 CFU per day
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare the effect of a probiotic strain on mental wellbeing in moderately stressed, healthy, adults in the general population. The main question it aims to answer is

• what is the impact of probiotic consumption on overall mental wellbeing? Participants will consume one probiotic or placebo capsule per day, answer a set of questionnaire (at 3 time points) and wear a wearable device for the total duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18-60 years old
* Currently living in the US.
* Have access to a smart phone, internet and computer.
* Report moderate levels of perceived stress.

Exclusion Criteria:

* Are currently taking medication for depression or anxiety
* Have had antibiotics within the previous month
* Have an allergy to coconut

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-09-16 (Actual); Study Completion 2023-09-16 (Actual)

PRIMARY OUTCOMES:
Change in Mental wellbeing | 4 weeks
  Improvement in mental wellbeing will be measured using the Oxford Happiness Questionnaire (OHQ).
  The Oxford Happiness Inventory was devised as a broad measure of personal happiness. The OHQ has a total of 29 items. Each item is scored on a Likert scale from 1 to 6 (1=strongly disagree; 2=moderately disagree; 3=slightly disagree; 4=slightly agree; 5=moderately agree; 6=strongly agree). Some items are phrased positively and others negatively. Such that negative items (1, 3, 12, 13, 16, 18, 21 and 29) should be scored in reverse (Hills & Argyle, 2002). The total score is then divided by 29. Interpretation of the final score is as follows: A final score between 1 to 2 is considered "not happy"; between 2 and 3 is "somewhat unhappy"; between 3 and 4 is considered "Neutral"; 4 is "somewhat or moderately happy"; between 4 and 5 is "rather happy"; between 5 and 6 is "very happy"; 6 is "too happy".

SECONDARY OUTCOMES:
Change in Stress scores | 4 weeks
  Change in stress scores will be measured using the short version of the Depression, Anxiety, Stress Scale (DASS-21). Each item is scored from 0 to 3, with a score of 0 indicating that the statement did not apply or never. A score of 3 indicates that the statement applied very much or almost always. In DASS-21, items 1, 6, 8, 11, 12, 14 and 18 relate to measurement of stress. Given that DASS-21 is the short version of DASS-42, the total item score is multiplied by 2. The final total scores range from 0 (no stress) to 42 (extremely stressed). Scores ranging between 0-14 (stress) are considered normal. Scores above 14 are considered positive for stress.
Change in anxiety scores | 4 weeks
  Change in anxiety scores will be measured using the short version of the Depression, Anxiety, Stress Scale (DASS-21). Each item is scored from 0 to 3, with a score of 0 indicating that the statement did not apply or never. A score of 3 indicates that the statement applied very much or almost always. In DASS-21, items 2, 4, 7, 9, 15, 19 and 20 relate to measurement of anxiety. Given that DASS-21 is the short version of DASS-42, the total item score is multiplied by 2. The final total scores range from 0 (no anxiety) to 42 (extremely anxious). Scores ranging between 0-14 (stress) are considered normal. Scores above 14 are considered positive for anxiety.
Change in Depression scores | 4 weeks
  Change in depression scores will be measured using the short version of the Depression, Anxiety, Stress Scale (DASS-21). Each item is scored from 0 to 3, with a score of 0 indicating that the statement did not apply or never. A score of 3 indicates that the statement applied very much or almost always. In DASS-21, items 3, 5, 10, 13, 16, 17, and 21 relate to measurement of depression . Given that DASS-21 is the short version of DASS-42, the total item score is multiplied by 2. The final total scores range from 0 (no depression ) to 42 (extremely depressed). Scores ranging between 0-14 (stress) are considered normal. Scores above 14 are considered positive for depression .
Change in Salivary cortisol | 4 weeks
  The saliva kit contains contains a 15 ml sterile plastic tube with lid and instructions. The instructions outline that the participant will need to self-collect the saliva sample before going to bed by spitting into the tube to fill up ½ of the tube. The collection process should take no more than 15-30 minutes total. The participant shall writ their name, the date, and the time of collection on the tube. The full sample volume will be used for measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Divya Nair, Principal Investigator — SunGenomics
Locations (1):
- Sun Genomics, Inc., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No